CLINICAL TRIAL: NCT00145392
Title: Body Composition, Glucose Metabolism, Insulin Resistance and Gene Expression in Muscle Cells in Healthy Overweight Women
Status: Completed | Type: Observational
Sponsor: Odense University Hospital (Other)
Responsible Party: Odense University Hospital
Other Study IDs: 005
Record Dates: First submitted 2005-09-02; First posted 2005-09-05 (Estimated); Last update posted 2008-06-24 (Estimated); Status verified 2008-06

CONDITIONS: Obesity; Type 2 Diabetes; Polycystic Ovary Syndrome
Keywords: Polycystic ovary syndrome; growth hormone; insulin resistance; overweight; glucose metabolism
MeSH Terms: conditions — Obesity; Diabetes Mellitus, Type 2; Polycystic Ovary Syndrome; Insulin Resistance; Overweight

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
In this study, we will clarify the degree of insulin resistance and characterise muscle glucose metabolism and gene expression in a group of overweight healthy women. The study will clarify how overweight influences body glucose metabolism and thereby in the long-run increases the risk for developing type 2 diabetes. Moreover, the study may clarify why some overweight women develop hormone disorders and diabetes while others remain healthy.

The study is essential as many patients suffer from diseases aggravated by overweight. In addition, a genetic disposition for diabetes or polycystic ovary syndrome may give rise to the disease if the patient gains weight. It is therefore important that weight-matched control subjects are included in projects with overweight patients.

This clinical trial includes 10 overweight women with regular hormones and normal level of male sex hormone. The patients included must be healthy, take no medications influencing the study results. The subjects must take no contraceptive pills or receive any other hormone treatment.

In connection with the investigation, the following will be carried out on all patients: clinical examination, blood tests, hyperinsulinaemic euglycaemic clamp, muscle biopsies, bone scan.

The purpose of the study is to gain more knowledge of how overweight influences women's risk of developing hormone diseases and diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Regular menses, i.e. cyclus length 25-34 days
* Premenopausal
* Ferrimann-Gallway score < 2
* BMI > 27 kg/m2
* normal total testosterone value < 3.5 nmol/l

Exclusion Criteria:

* Age <18 years
* Contraceptive pills within the past 3 months
* Postmenopausal (increased FSH)
* Diabetes mellitus
* Endocrine or other disease requiring treatment
* Eating disorder or other psychiatric history
* Drug use known to influence parameters investigated in this trial
* Pregnancy

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10
Dates: Start 2002-09; Primary Completion 2007-01 (Actual); Study Completion 2007-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dorte Glintborg, MD, Principal Investigator — Odense University Hospital
Locations (1):
- Department of Endocrinology, Odense University Hospital, Odense, Funen, Denmark